CLINICAL TRIAL: NCT00334334
Title: To Assess Safety, Reactogenicity and Immunogenicity of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine, When Co-administered With DTPa-combined Vaccines and MenC or Hib-MenC Vaccines During the First 6 Months of Age.
Brief Title: Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' 10-valent Pneumococcal Conjugate Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107005
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus pneumonia, vaccine
MeSH Terms: conditions — Streptococcal Infections; Pneumonia | interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Three dose primary vaccination of healthy infants between 6 to 16 weeks of age at the time of the first vaccination against Streptococcus pneumonia, Neisseria meningitidis and Haemophilus influenzae type b.

ELIGIBILITY:
Inclusion Criteria:

* male or female between, and including, 6-16 weeks (42 to 118 days) of age at the time of the first vaccination, free of obvious health problems and with written informed consent obtained from the parent/guardian of the subject.

Exclusion Criteria:

* use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the entire study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before each dose of vaccine(s) and ending 7 days after dose 1 and dose 2 or 1 month after dose 3.
* Previous vaccinations against diseases which are targeted by the vaccines used in the study.

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1572 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Post at least 1 dose: rectal fever >39°C

SECONDARY OUTCOMES:
Post each dose: solicited/unsolicited AEs (4/31 days), SAEs (whole study); post dose 2 & 3: Ab conc to vaccine antigens

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (56):
- Germany (37):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Roding, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Niedernhausen, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Herford, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Bodenheim, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gerolstein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Singwitz, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Weimar, Thuringia
- Poland (7):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Wola
- Spain (12):
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Montgat/Barcelona
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, San T Vicenç Del Horts ( Barcelona)
  - GSK Investigational Site, Tona/Barcelona
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vélez-Málaga / Málaga

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chevallier B, Vesikari T, Brzostek J, Knuf M, Bermal N, Aristegui J, Borys D, Cleerbout J, Lommel P, Schuerman L. Safety and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with routine childhood vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S109-18. doi: 10.1097/INF.0b013e318199f62d. PMID 19325447
- [Background] Hausdorff WP, Dagan R, Beckers F, Schuerman L. Estimating the direct impact of new conjugate vaccines against invasive pneumococcal disease. Vaccine. 2009 Dec 9;27(52):7257-69. doi: 10.1016/j.vaccine.2009.09.111. Epub 2009 Oct 13. PMID 19833248
- [Background] Hausdorff WP et al. Estimation of the direct impact of a 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHID-CV) candidate against invasive pneumococcal disease (IPD). Abstract presented at the 6th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD), Reykjavik, Iceland, 8-12 June 2008.
- [Background] Knuf M, Szenborn L, Moro M, Petit C, Bermal N, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of routinely used childhood vaccines when coadministered with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S97-S108. doi: 10.1097/INF.0b013e318199f61b. PMID 19325452
- [Background] Knuf M et al. Safety and reactogenicity of the new 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHID-CV). Abstract presented at the 6th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD), Reykjavik, Iceland, 8-12 June 2008.
- [Background] Poolman J, Frasch C, Nurkka A, Kayhty H, Biemans R, Schuerman L. Impact of the conjugation method on the immunogenicity of Streptococcus pneumoniae serotype 19F polysaccharide in conjugate vaccines. Clin Vaccine Immunol. 2011 Feb;18(2):327-36. doi: 10.1128/CVI.00402-10. Epub 2010 Dec 1. PMID 21123523
- [Background] Poolman J et al. Anti-pneumococcal serotype 19F/A antibody functionality is influenced by the vaccine conjugation method. Abstract presented at the PHAA, 12th National Immunisation Conference. Adelaide, Australia, 17-19 August 2010.
- [Background] Poolman J et al. Functionality of conjugate vaccine-induced antibodies against pneumococcal serotype 19F is influenced by the conjugation method. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L, Borys D, Hoet B, Forsgren A, Prymula R. Prevention of otitis media: now a reality? Vaccine. 2009 Sep 25;27(42):5748-54. doi: 10.1016/j.vaccine.2009.07.070. Epub 2009 Aug 8. PMID 19666154
- [Background] Schuerman L, Wysocki J, Tejedor JC, Knuf M, Kim KH, Poolman J. Prediction of pneumococcal conjugate vaccine effectiveness against invasive pneumococcal disease using opsonophagocytic activity and antibody concentrations determined by enzyme-linked immunosorbent assay with 22F adsorption. Clin Vaccine Immunol. 2011 Dec;18(12):2161-7. doi: 10.1128/CVI.05313-11. Epub 2011 Oct 12. PMID 21994351
- [Background] Schuerman L et al. Immune responses against cross-reactive pneumococcal serotypes 6A and 19A with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Immune responses to the non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) appear not influenced by co-administration with DTPw-combination vaccine. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. OPA assay is more reliable predictor of vaccine effectiveness against invasive pneumococcal disease (IPD) than ELISA antibody measurements. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Population variability in antibody responses following pneumococcal conjugate vaccination: experience with the non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Population variability of opsonophagocytic activity following 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate (PHiD-CV) vaccination more limited than antibody responses. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Prevention of invasive pneumococcal disease and meningitis with PHiD-CV when used according to a 2+1 schedule. Abstract presented at the Meningitis Research Foundation Conference (MRFC). London, UK, 11-12 November 2009.
- [Background] Tejedor JC et al. Co-administration of the new 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHIDCV) with other routine paediatric vaccines. Abstract presented at the 6th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD), Reykjavik, Iceland, 8-12 June 2008.
- [Background] Vesikari T, Wysocki J, Chevallier B, Karvonen A, Czajka H, Arsene JP, Lommel P, Dieussaert I, Schuerman L. Immunogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) compared to the licensed 7vCRM vaccine. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S66-76. doi: 10.1097/INF.0b013e318199f8ef. PMID 19325449
- [Background] Wysocki J, Tejedor JC, Grunert D, Konior R, Garcia-Sicilia J, Knuf M, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with different neisseria meningitidis serogroup C conjugate vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S77-88. doi: 10.1097/INF.0b013e318199f609. PMID 19325450
- [Background] Wysocki J et al. Immunogenicity of the new 10-valent pneumoccocal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHiDCV) in infants after 3-dose priming before 6 months of age. Abstract presented at the 6th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD), Reykjavik, Iceland, 8-12 June 2008.
- [Derived] Tejedor JC, Brzostek J, Konior R, Grunert D, Kolhe D, Baine Y, Van Der Wielen M. Antibody Persistence in Young Children 5 Years after Vaccination with a Combined Haemophilus influenzae Type b-Neisseria meningitidis Serogroup C Conjugate Vaccine Coadministered with Diphtheria-Tetanus-Acellular Pertussis-Based and Pneumococcal Conjugate Vaccines. Clin Vaccine Immunol. 2016 Jul 5;23(7):555-63. doi: 10.1128/CVI.00057-16. Print 2016 Jul. PMID 27145999
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 107005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register